CLINICAL TRIAL: NCT01222793
Title: Effects of Antipsychotics on Eating and Food Craving in People With Schizophrenia
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910460; 10-DA-N460
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-05-03

CONDITIONS: Schizophrenia; Obesity
Keywords: High Weight Gain Liability (HWLA); Antipsychotic; Obesity; Low Weight Gain; Schizophrenia; Food Craving
MeSH Terms: conditions — Schizophrenia; Obesity; Weight Gain

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Although second-generation antipsychotic medications have fewer serious side effects and complications than first-generation ones, they are strongly associated with weight gain for reasons that are as yet unknown. Comparing the effects of second-generation antipsychotics with a high weight-gain liability (HWGL) low weight-gain liability (LWGL) antipsychotics may provide more information on which medications are best suited for different individuals. Researchers are interested in studying how people taking various antipsychotics compare with controls in regard to food craving and eating behavior. This knowledge should help to guide practitioners when advising patients about the weight-gain effects of these medications.

Objectives:

- To examine eating behavior and food craving in patients with schizophrenia who are taking HWGL antipsychotics compared with those taking LWGL antipsychotics and with healthy controls taking no antipsychotics.

Eligibility:

* Individuals between 18 and 45 years of age who have been diagnosed with schizophrenia or a related disorder, have a body mass index between 25 and 29.9, and have never had an eating disorder.
* Healthy individuals between 18 and 45 years of age who have a body mass index between 25 and 29.9 and have never had an eating disorder.

Design:

* This study involves an initial screening visit and four study visits.
* Participants will be screened with a medical history and physical examination, as well as questionnaires about stress levels, food cravings, smoking, exercise, and eating habits; a taste test; and saliva collection (to measure stress hormones).
* Visit 2: Participants will have an optional overnight stay, and will provide blood samples before having a breakfast beverage and answering questions about tiredness, anxiety, hunger, and alertness during a 1.5 hour session.

Visit 3: Participants will have an optional overnight stay and a light breakfast, followed by blood draws and questions about hunger and food cravings.

Visit 4: Participants will have an optional overnight stay, followed by questions about food preference. Participants will not be allowed to eat until mid-morning of the next day.

Visit 5: Participants will eat normally before arriving at the research site, and will have tests to measure food craving and questionnaires about mood and feelings.

DETAILED DESCRIPTION:
Objective

Some second-generation antipsychotics, such as olanzapine and clozapine, seem especially prone to induce metabolic complications and substantial increases in weight. The mechanisms of these side effects are unknown, but may include antagonism at histamine H1 receptors. We will refer to olanzapine and clozapine as antipsychotics with a high weight-gain liability (HWGL). The primary aim of this project is to examine eating and food craving in patients with schizophrenia who are taking HWGL antipsychotics compared with those taking LWGL antipsychotics (mid- to high-potency first-generation antipsychotics, aripiprazole, or ziparasidone) and compared with healthy controls taking no antipsychotics. The antipsychotics we are classifying as LWGL group do not have appreciable H1 receptor antagonism. We will exclude participants taking antipsychotics that have middling degrees of H1 receptor antagonism (e.g. quetiapine).

This study will help us understand how people with schizophrenia differ from controls on eating and food craving, as well as the effects of different classes of antipsychotics. This knowledge should help to guide practitioners when advising patients about the weight-gain effects of these medications. For example, if we find that participants on HWGL antipsychotics tend to crave high-fat foods, practitioners can work with patients to anticipate and mitigate this side effect.

Study population. The study population will be in- or outpatients with a DSM-IV diagnosis of schizophrenia or schizoaffective disorder stabilized on either olanzapine or clozapine (HWGL antipsychotics) (N=20), aripiprazole, ziprasidone, or a first-generation antipsychotic (LWGL antipsychotics) (n=20), and normal controls (people with no Axis I psychiatric disorder taking no antipsychotic medication) (n=20), for a total of 60 participants. All participants will be between the ages of 18 to 45 years and considered overweight (BMI greater than or equal to 25 and less than or equal to 29.9 kg/m(SqrRoot)). The pediatric population has been excluded to rule out certain hormonal effects (e.g. puberty) on eating behavior. A BMI range encompassing participants that are overweight was selected to maximize recruitment and to minimize confounding effects of BMI on eating behavior. Exclusion criteria will include weight-related conditions and current dietary restrictions.

Experimental design and methods. In a between-subjects design, the three study groups will be compared in terms of four domains of eating behavior: (1) food craving, (2) satiety signaling, (3) meal size (satiation), and (4) food preferences. Assessments will occur during five study visits (including an initial visit for consenting and screening).

Outcome measures: Primary outcome measures will include a preload-test meal paradigm (satiety), meal size perception and satiation, food preference, food craving, and gustatory functioning. Secondary measures will include: Weight and Eating Assessment questionnaire, Recent Physical Activity Questionnaire (RPAQ), State Trait Anxiety Inventory (STAI), Exercise Motivations Inventory (EMI), Childhood Trauma Questionnaire, Tobacco Craving Questionnaire-Short Form (TCQ-SF), Fagerstrom Test for Nicotine Dependence (FTND), BMI, hip/waist measurements, and fasting blood work: CBC, CMP14, lipid panel, leptin, ghrelin, adiponectin, and thyroid panel.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants must:

* be between age 18 and 45.
* have a BMI between 25 or above.

Participants in the antipsychotic-medication groups must:

1. meet DSM-IV criteria for schizophrenia or schizoaffective disorder, and have been stabilized on an antipsychotic medication for the past 3 months. Antipsychotics include olanzapine, clozapine, aripiprazole, ziprasidone, and first-generation antipsychotics (mid to high potency). Polypharmacy is allowed as long as both medications fit into the same grouping (HWGL or LWGL).

Healthy controls must:

1. have no DSM IV Axis I disorder (Schizophrenia or schizoaffective disorder, Depression, Bipolar Disorder) based on a SCID interview.

EXCLUSION CRITERIA:

Participants will be excluded if they:

meet DSM-IV criteria for a past and/or current eating disorder via the SCID, or if they have a past medical history of an eating disorder, received treatment/counseling for an eating disorder and/or required hospitalization for an eating disorder. (If an otherwise undiagnosed eating disorder is detected during screening, referral to treatment will be provided.)

are taking risperidone, quetiapine, paliperidone, iloperidone, or low-potency first-generation antipsychotics (see Appendix A for complete list of excluded medications).

are taking weight-loss medications, whether over-the-counter (i.e. Hydroxycut, Stacker products, Metabo-Plus, CortiSlim), or prescribed, including appetite suppressants (Didrex, Tenuate, Sanorex, Mazanor, Adipex-P, Meridia, and Phentermine) and fat-absorption inhibitors (Xenical).

are currently enrolled in a nutrition-based weight-loss program (i.e. Weight Watchers, Jenny Craig, Nutri-System).

have undergone weight-loss surgery (i.e. banding, gastric bypass surgery, sleeve gastrectomy, liposuction).

have Cushing's syndrome, polycystic-ovary syndrome, hyperthyroidism, hypothyroidism, or a DSM-IV diagnosis of depression.

have Type I or Type II diabetes, defined as a fasting blood glucose level of greater than or equal to 99.

have cognitive impairment severe enough to preclude informed consent or valid responses on questionnaires. This is defined an as a score of less than 10 on the Evaluation to Sign Consent (ESC) and judged by the treating clinician. Participants obtaining a 10 on the ESC are re-briefed on the item that they missed, and are asked the question again until they get it correct to ensure their understanding.

have a medical illness that, in the view of the investigators, would compromise participation.

have dietary restrictions or food allergies that, in the view of the investigators, would compromise participation.

are pregnant (as this might alter appetite or cravings).

have begun or stopped smoking in the previous 3 months

Also, participants will be excluded from the control group if they:

are taking antipsychotics, antidepressants or mood stabilizers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09-26; Study Completion 2012-05-03

CONTACTS AND LOCATIONS:
Overall Officials: Carol Myers, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Background] Addington D, Addington J, Maticka-Tyndale E. Assessing depression in schizophrenia: the Calgary Depression Scale. Br J Psychiatry Suppl. 1993 Dec;(22):39-44. PMID 8110442
- [Background] Andreasen NC. Negative symptoms in schizophrenia. Definition and reliability. Arch Gen Psychiatry. 1982 Jul;39(7):784-8. doi: 10.1001/archpsyc.1982.04290070020005. PMID 7165477
- [Background] Baptista T, De Mendoza S, Beaulieu S, Bermudez A, Martinez M. The metabolic syndrome during atypical antipsychotic drug treatment: mechanisms and management. Metab Syndr Relat Disord. 2004 Fall;2(4):290-307. doi: 10.1089/met.2004.2.290. PMID 18370698